CLINICAL TRIAL: NCT01594931
Title: A Randomised, Multi-Centre, Phase II, Dose-ranging Clinical Study to Assess the Safety and Efficacy of Fixed Dose, Orally Administered Pyronaridine and Artesunate (3:1) in Adult Patients With Acute Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Phase II Dose-ranging Study of Pyronaridine/Artesunate in Adults Patients With Plasmodium Falciparum Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP-C-002-05
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Results first posted 2021-09-17 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: malaria; antimalarial; artemisinin based combination therapy (ACT); pyronaridine artesunate (Pyramax)
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- pyronaridine/artesunate (6:2 mg/kg) (Experimental): pyronaridine tetraphosphate 6 mg/kg and artesunate 2 mg/kg
  Interventions: Drug: pyronaridine/artesunate
- pyronaridine/artesunate (9:3 mg/kg) (Experimental): pyronaridine tetraphosphate 9 mg/kg and artesunate 3 mg/kg
  Interventions: Drug: pyronaridine/artesunate
- pyronaridine/artesunate (12:4 mg/kg) (Experimental): pyronaridine tetraphsophate 12 mg/kg and artesunate 4 mg/kg
  Interventions: Drug: pyronaridine/artesunate

INTERVENTIONS:
Drug: pyronaridine/artesunate — Tablets of fixed dose combination of pyronaridine and artesunate at a ratio of 3:1. The tablets were taken daily for 3 days.
  Other Names: Pyramax

SUMMARY:
The primary trial objective is to determine the clinically effective dose of orally administered pyronaridine/artesunate (Pyramax®, PA) with a 3:1 ratio to treat adults with acute, symptomatic, uncomplicated P. falciparum malaria in South East Asia and Africa. Secondary trial objectives are to determine the safety of once-daily dosing for 3 days of PA and to explore possible ethnic differences in safety or efficacy.

DETAILED DESCRIPTION:
This is a double-blind, multicentre, randomized, parallel group, dose-finding study of the efficacy, safety and tolerability of a once-daily 3-day regimen of PA with a 3:1 weight/weight ratio for patients with acute, symptomatic, uncomplicated P. falciparum malaria. Patients will be recruited from 5 to 7 study sites in endemic regions of South East Asia and Africa and will be randomized to 1 of 3 treatment groups differing in dosage, with 160 patients per group (n-480). Randomization will be balanced within each study site across all 3 study groups in pre-assigned treatment blocks.

The first dose will be administered on Day 0 and patients will remain hospitalized for at least 4 days whilst undertaking the 3-day regimen. Patients will remain near the study site for a minimum of 7 days or once fever and parasite clearance is confirmed (assessed by 3 negative readings of fever and/or slide).

The primary efficacy end point is the cure rate on Day 28 - the proportion of patients with PCR-corrected adequate clinical and parasitological response (ACPR). Despite this Day 28 end point, the relatively long half-life of pyronaridine necessitates follow-up until Day 42. In the case of adverse events reported and unresolved at Day 42, patients will be followed up for a further 30 days, or until resolution of the event.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between the age of 15 and 60 years of age inclusive
2. Written informed consent, in accordance with local practice, provided by patient and/or parent/guardian/spouse. If the patient is unable to write, witnessed consent is permitted according to local ethical considerations
3. Absence of severe malnutrition (defined as the weight-for-height being below -3 standard deviations or <70% of the median of the NCHS/WHO normalized reference values)
4. Weight of between 35 kg and 75 kg inclusive
5. Presence of acute symptomatic uncomplicated P. falciparum malaria with a diagnosis confirmed by a positive blood smear with asexual forms of P. falciparum only (i.e. no mixed infection) plus history of fever within the previous 24 hours or a measured temperature of ≥37.5°C (depending on method of measurement):

   * the acceptable range is between 1,000 and 100,000 asexual parasite count/μl of blood and
   * axillary/tympanic temperature of ≥ 37.5°C or oral/rectal temperature of ≥ 38.0°C
6. Ability to swallow oral medication
7. Ability to comply with study visit schedule: patients will be hospitalised for at least 4 days and will be required to remain in the vicinity of the trial site for a minimum of 7 days or until clearance of fever and parasite for at least 24 hours, whichever is the later. The patient is to return to the study site or to make themselves available for all scheduled follow up visits, until discharge at Day 42.
8. Females must not be pregnant or lactating and be willing to take measures to not become pregnant during the study period
9. Willingness and ability to comply with the study protocol for the duration of the study

Exclusion Criteria:

1. Patients with signs and symptoms of severe/complicated malaria requiring parenteral treatment according to the World Health Organization Criteria 2000
2. Mixed Plasmodium infection
3. Severe vomiting, defined as >3 times in the 24 hours prior to inclusion in the trial or inability to tolerate oral treatment
4. Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia), respiratory (including active tuberculosis), hepatic, renal, gastrointestinal, immunological (including active HIV-AIDS), neurological (including auditory), endocrine, infectious, malignancy, psychiatric or other clinically important abnormality (including head trauma).
5. Presence of febrile conditions caused by diseases other than malaria
6. Known history of hypersensitivity, allergic or adverse reactions to pyronaridine or artesunate or other artemisinins
7. Evidence of use of any other antimalarial agent within 2 weeks prior to the start of the study confirmed by a negative urine test or using Eggelte dipsticks
8. Positive urine pregnancy test or lactating
9. Received an investigational drug within the past 4 weeks
10. Known active Hepatitis A IgM (HAV-IgM), Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV Ab)
11. Known seropositive HIV antibody
12. Liver function tests [ASAT/ALAT levels] >2.5 times upper limit of normal values
13. Known significant renal impairment as indicated by a serum creatinine of ≥ 1.4 mg/dl
14. Previous participation in this clinical trial

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 477 (Actual)
Dates: Start 2005-07; Primary Completion 2006-03 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sornchai Looareesuwan, MD, Principal Investigator — Hospital of Tropical Diseases, Mahidol University, Bangkok, Thailand; Duong Socheat, MD, Principal Investigator — Nat. Centre for Parasitol., Entomol. and Malaria Control, Phnom Penh, Cambodia; Emiliana Tjitra, PhD, Principal Investigator — Bethesda Hospital, Tomohon, North Sulawasi, Indonesia; Kalifa Bojang, MD, Principal Investigator — MRC Laboratories, Faraffeni, The Gambia; Patrice Piola, MD, Principal Investigator — Epicentre, Mbarara, Uganda; Oumar Gaye, MD, Principal Investigator — Centre de santé Roi Baudouin, Guediawaye, Senegal
Locations (6):
- Pailin General Hospital, Pailin, Cambodia
- Bethesday Hospital, Tomohon, North Sulawesi, Indonesia
- Centre de santé du roi Baudoin, Guédiawaye, Senegal
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand
- Farafenni Field Station, c/o MRC Laboratories, Farafenni, The Gambia
- MSF Epicentre, Mbarara, Uganda

REFERENCES:
- [Derived] Duparc S, Borghini-Fuhrer I, Craft CJ, Arbe-Barnes S, Miller RM, Shin CS, Fleckenstein L. Safety and efficacy of pyronaridine-artesunate in uncomplicated acute malaria: an integrated analysis of individual patient data from six randomized clinical trials. Malar J. 2013 Feb 21;12:70. doi: 10.1186/1475-2875-12-70. PMID 23433102

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Pyronaridine/Artesunate (6:2 mg/kg): Pyronaridine tetraphosphate 6 mg/kg and artesunate 2 mg/kg
  Pyronaridine/artesunate: Tablets of fixed dose combination of pyronaridine and artesunate at a ratio of 3:1
- Group B: Pyronaridine/Artesunate (9:3 mg/kg): Pyronaridine tetraphosphate 9 mg/kg and artesunate 3 mg/kg
  Pyronaridine/artesunate: Tablets of fixed dose combination of pyronaridine and artesunate at a ratio of 3:1
- Group C: Pyronaridine/Artesunate (12:4 mg/kg): Pyronaridine tetraphsophate 12 mg/kg and artesunate 4 mg/kg
  Pyronaridine/artesunate: Tablets of fixed dose combination of pyronaridine and artesunate at a ratio of 3:1
Period: Overall Study
Arm/Group | Group A: Pyronaridine/Artesunate (6:2 mg/kg) | Group B: Pyronaridine/Artesunate (9:3 mg/kg) | Group C: Pyronaridine/Artesunate (12:4 mg/kg)
Started | 160 | 157 | 160 (One randomized subject was not treated.)
Completed | 131 | 145 | 146
Not Completed | 29 | 12 | 14
Not completed — Adverse Event | 3 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1
Not completed — Lack of Efficacy | 7 | 2 | 2
Not completed — Lost to Follow-up | 4 | 3 | 3
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — No defiined | 11 | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Pyronaridine/Artesunate (6:2 mg/kg) | Group B: Pyronaridine/Artesunate (9:3 mg/kg) | Group C: Pyronaridine/Artesunate (12:4 mg/kg) | Total
Number analyzed (Participants) | 160 | 157 | 160 | 477
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One subject, who was randomized to the 12+4 mg/kg dose group, did not receive any study medication and was excluded from all populations.
  years
    number analyzed (Participants) | 160 | 157 | 159 | 476
    (all) | 27.0 (10.9) | 27.4 (10.9) | 28.9 (11.4) | 27.8 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject, who was randomized to the 12+4 mg/kg dose group, did not receive any study medication and was excluded from all populations.
  Participants
    number analyzed (Participants) | 160 | 157 | 159 | 476
    Female | 43 | 37 | 40 | 120
    Male | 117 | 120 | 119 | 356
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One subject, who was randomized to the 12+4 mg/kg dose group, did not receive any study medication and was excluded from all populations.
  Participants
    number analyzed (Participants) | 160 | 157 | 159 | 476
    White/Caucasian | 0 | 0 | 0 | 0
    Black | 49 | 47 | 48 | 144
    Asian/Oriental | 111 | 110 | 111 | 332
Region of Enrollment [Number; unit: participants]
  Cambodia | 10 | 9 | 10 | 29
  Senegal | 32 | 32 | 30 | 94
  Gambia | 12 | 10 | 13 | 35
  Uganda | 5 | 5 | 6 | 16
  Thailand | 80 | 80 | 80 | 160
  Indonesia | 21 | 21 | 21 | 63

OUTCOME MEASURES:

1. Primary Outcome: PCR-Corrected ACPR at Day 28
Description: Percentage of subjects with PCR-corrected adequate clinical and parasitological response (ACPR) on Day 28, defined as absence of parasitaemia on Day 28 without the subject's meeting any of the criteria of early treatment failure, late clinical failure, or late parasitological failure
Time Frame: Day 28
Population: Subjects meeting the following: completed a full course of study medication and had known efficacy endpoints; no missed dose due to vomiting (except at D0); no concom. medication, except acetaminophen; no concom. disease that could have interfered with treatment outcome; no major protocol violation with respect to entry eligibility criteria.
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Group A: Pyronaridine/Artesunate (6:2 mg/kg) | Group B: Pyronaridine/Artesunate (9:3 mg/kg) | Group C: Pyronaridine/Artesunate (12:4 mg/kg)
Number analyzed (Participants) | 101 | 103 | 102
percentage of subjects | 95 [89.9 to 98.0] | 99 [95.5 to 100.0] | 99 [95.4 to 99.9]

2. Secondary Outcome: PCR-Corrected ACPR at Day 14
Description: Percentage of subjects with PCR-corrected adequate clinical and parasitological response (ACPR) on Day 14, defined as absence of parasitaemia on Day 14 without the subject's meeting any of the criteria of early treatment failure, late clinical failure, or late parasitological failure
Time Frame: Day 14
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of subjects
Arm/Group | Group A: Pyronaridine/Artesunate (6:2 mg/kg) | Group B: Pyronaridine/Artesunate (9:3 mg/kg) | Group C: Pyronaridine/Artesunate (12:4 mg/kg)
Number analyzed (Participants) | 105 | 107 | 106
percentage of subjects | 100 [97.2 to 100.0] | 100 [97.2 to 100.0] | 100 [97.2 to 100.0]

3. Secondary Outcome: Parasite Clearance Time
Description: Parasite clearance time was defined as the time (in hours) from first dosing to the time of first blood draw with parasite clearance. Parasite clearance is defined as zero presence of parasites for two consecutive negative readings eight hours apart, with confirmed negative reading at 24 hours after the first negative slide
Time Frame: Thick blood slides were examined every 8 hours until at least 72 hours or until a negative smear was recorded
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group A: Pyronaridine/Artesunate (6:2 mg/kg) | Group B: Pyronaridine/Artesunate (9:3 mg/kg) | Group C: Pyronaridine/Artesunate (12:4 mg/kg)
Number analyzed (Participants) | 108 | 109 | 109
hours | 36.9 (20.73) | 33.6 (17.08) | 30.8 (14.96)

4. Secondary Outcome: Fever Clearance Time
Description: Fever clearance time was defined as the time (in hours) from first dosing to the first normal reading with fever clearance (2 consecutive assessments without fever (<37.5°C)). The method of temperature measurement was the same (ie, axillary, tympanic, oral or rectal) for each subject. Any subjects with a documented history of fever at inclusion, but who did not subsequently have a documented temperature reading >37.5°C during the 24 hours after initial dosing, were not included in this end point analysis.
Time Frame: Every 8 hours for at least 72 hours after the first dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group A: Pyronaridine/Artesunate (6:2 mg/kg) | Group B: Pyronaridine/Artesunate (9:3 mg/kg) | Group C: Pyronaridine/Artesunate (12:4 mg/kg)
Number analyzed (Participants) | 84 | 93 | 93
hours | 16.8 (12.75) | 24.0 (25.99) | 17.0 (12.90)

5. Secondary Outcome: Parasite Clearance
Description: Parasite clearance is defined as zero presence of parasites for 2 consecutive negative readings 8 hours apart, with confirmed negative reading at 24 hours after the first negative slide. The proportion of subjects with parasite clearance was summarized at Days 1, 2, and 3.
Time Frame: Days 1, 2, and 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group A: Pyronaridine/Artesunate (6:2 mg/kg) | Group B: Pyronaridine/Artesunate (9:3 mg/kg) | Group C: Pyronaridine/Artesunate (12:4 mg/kg)
Number analyzed (Participants) | 108 | 109 | 109
percentage of subjects
  Clearance rate (%) at Day 1 (24h after first dose) | 74 [64.8 to 82.0] | 82 [73.1 to 88.4] | 84 [76.2 to 90.6]
  Clearance rate (%) at Day 2 (48h after first dose) | 93 [85.9 to 96.7] | 96 [90.9 to 99.0] | 95 [89.6 to 98.5]
  Clearance rate (%) at Day 3 (72h after first dose) | 96 [90.8 to 99.0] | 98 [93.5 to 99.8] | 99 [95.0 to 100.0]

6. Secondary Outcome: Fever Clearance
Description: Fever clearance was defined as a subject without fever for 2 consecutive assessments, plus confirmed normal temperature at 24 hours. The proportion of subjects with fever clearance was summarized at Days 1, 2, and 3.
Time Frame: Days 1, 2 and 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group A: Pyronaridine/Artesunate (6:2 mg/kg) | Group B: Pyronaridine/Artesunate (9:3 mg/kg) | Group C: Pyronaridine/Artesunate (12:4 mg/kg)
Number analyzed (Participants) | 108 | 109 | 109
percentage of subjects
  Clearance rate (%) at Day 1 (24h after first dose) | 96 [90.8 to 99.0] | 91 [83.8 to 95.5] | 96 [90.9 to 99.0]
  Clearance rate (%) at Day 2 (48h after first dose) | 99 [94.9 to 100.0] | 96 [90.9 to 99.0] | 100 [96.7 to 100.0]
  Clearance rate (%) at Day 3 (72h after first dose) | 99 [94.9 to 100.0] | 96 [90.9 to 99.0] | 100 [96.7 to 100.0]

7. Secondary Outcome: Adverse Events (AEs)
Description: An AE was defined as any unfavourable and unintended sign, symptom, syndrome, or illness that developed or worsened during the period of observation in the clinical study
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study or resolution of the event, whichever was earlier
Population: The safety population includes all subjects who were randomized and received any study medication, regardless of the amount.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A: Pyronaridine/Artesunate (6:2 mg/kg) | Group B: Pyronaridine/Artesunate (9:3 mg/kg) | Group C: Pyronaridine/Artesunate (12:4 mg/kg)
Number analyzed (Participants) | 160 | 157 | 159
Participants
  Nr subj. with ≥1 AE | 106 | 90 | 91
  Nr subj. with ≥1 treatment-related AE | 35 | 33 | 36
  Nr subj. with ≥1 SAE | 3 | 0 | 1
  Nr subj. with ≥1 treatment-related SAE | 0 | 0 | 1
  Nr subj. with ≥1 AE leading to death | 0 | 0 | 0
  Nr subj. with ≥1 AE leading to study withdrawal | 3 | 1 | 1

ADVERSE EVENTS:
Time Frame: Day 0 to 42. Subjects experiencing AEs at Day 42 were followed for up to 30 days after the end of study or resolution of the event, whichever was earlier
Arm/Group | Group A: Pyronaridine/Artesunate (6:2 mg/kg) | Group B: Pyronaridine/Artesunate (9:3 mg/kg) | Group C: Pyronaridine/Artesunate (12:4 mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/157 | 0/159
Serious Adverse Events (participants affected / at risk) | 3/160 | 0/157 | 1/159
Other Adverse Events (participants affected / at risk) | 106/160 | 90/157 | 91/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Pyronaridine/Artesunate (6:2 mg/kg) (N=160) | Group B: Pyronaridine/Artesunate (9:3 mg/kg) (N=157) | Group C: Pyronaridine/Artesunate (12:4 mg/kg) (N=159)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A: Pyronaridine/Artesunate (6:2 mg/kg) (N=160) | Group B: Pyronaridine/Artesunate (9:3 mg/kg) (N=157) | Group C: Pyronaridine/Artesunate (12:4 mg/kg) (N=159)
Anaemia (Blood and lymphatic system disorders) | 16 (16) | 15 (15) | 13 (13)
Eosinophilia (Blood and lymphatic system disorders) | 6 (6) | 7 (7) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 10 (10) | 7 (9) | 8 (8)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 6 (6) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 4 (4) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 3 (4)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (12) | 8 (8) | 8 (9)
Asthenia (General disorders) | 2 (2) | 4 (4) | 0 (0)
Chest pain (General disorders) | 0 (0) | 3 (3) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 1 (1)
Fatigue (Congenital, familial and genetic disorders) | 3 (3) | 4 (5) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Malaria (Infections and infestations) | 12 (12) | 8 (8) | 7 (7)
Nasopharyngitis (Infections and infestations) | 2 (2) | 3 (4) | 3 (3)
Otitis media acute (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Parasitic infection intestinal (Infections and infestations) | 4 (4) | 2 (2) | 4 (4)
Plasmodium falciparum infection (Infections and infestations) | 6 (6) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 4 (4) | 7 (8)
Alanine aminotransferase increased (Investigations) | 4 (4) | 6 (6) | 6 (6)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Eosinophil count increased (Investigations) | 17 (18) | 14 (15) | 14 (14)
Transaminases increased (Investigations) | 4 (4) | 3 (3) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (10) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 22 (24) | 19 (21) | 17 (18)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3) | 2 (2) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 7 (7) | 13 (14)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Rash (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No